CLINICAL TRIAL: NCT00006275
Title: Study of Topical Calcitriol in Children With Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Boston University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15372; BUSM-90-106
Record Dates: First submitted 2000-09-11; First posted 2000-09-12 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-09

CONDITIONS: Psoriasis
Keywords: dermatologic disorders; psoriasis; rare disease
MeSH Terms: conditions — Psoriasis; Skin Diseases; Rare Diseases | interventions — Calcitriol

INTERVENTIONS:
Drug: calcitriol

SUMMARY:
OBJECTIVES:

I. Determine the therapeutic efficacy and safety of topical calcitriol in children with psoriasis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients apply topical calcitriol in petrolatum on a psoriatic lesion daily. Patients also apply petrolatum without calcitriol to another psoriatic lesion daily.

Patients have both lesions photographed prior to therapy, monthly during therapy, and at the completion of therapy. Lesions are assessed weekly for 1 month and then every 2 weeks while on study. Blood samples are collected every 1 to 2 months and urine samples are collected every 2 weeks while on study.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of psoriasis At least 2 lesions with area at least 30-50 cm2

--Prior/Concurrent Therapy--

No other concurrent therapy for psoriasis No concurrent calcium supplements greater than 1,000 mg/day No concurrent prednisone or other drugs affecting serum or urine calcium levels

--Patient Characteristics--

Renal: No high blood or urinary calcium levels

Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 2000-07; Study Completion 2000-07

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. Holick, Study Chair — Boston University